CLINICAL TRIAL: NCT05178706
Title: Does the Upper Extremity Rehabilitation Program Implemented on Individuals With Facioscapulohumeral Dystrophy, Followed by Various Interventions, Have an Impact on Function, Balance, and Gait?
Brief Title: Effectiveness of Upper Extremity Rehabilitation in pwFSHD (Patient With Facioscapulohumeral Dystrophia)
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aysenur Erekdag, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: 60260273-615.98-
Record Dates: First submitted 2021-11-20; First posted 2022-01-05 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Facioscapulohumeral Muscular Dystrophy
Keywords: Neuromuscular Disease; Scapulothoracic Arthrodesis; Exercise Therapy; Kinetic Chain
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- non-operative conservative treatment: 9 individuals diagnosed with FSHD who have not undergone unilateral or bilateral surgery who meet the inclusion criteria.
  application of determined outcome scales and rehabilitation program on patients
  Interventions: Other: upper extremity rehabilitation program; Diagnostic Test: Results of assessment
- scapulothoracic arthrodesis: 9 individuals diagnosed with FSHD who have undergone bilateral surgery who meet the inclusion criteria.
  application of determined outcome scales and rehabilitation program on patients
  Interventions: Other: upper extremity rehabilitation program; Diagnostic Test: Results of assessment
- healthy control: 18 participants for measuring the normative datas; application of determined outcome scales
  Interventions: Diagnostic Test: Results of assessment

INTERVENTIONS:
Other: upper extremity rehabilitation program — Patients with FSHD who have undergone and have not undergone surgery will be given activity training by the same physiotherapist after they agree to participate in the study. Both groups will be given the same exercises, the same number of repetitions and the same frequency. A two-phase exercise protocol will be established and progression will be performed after 4 weeks. The exercises will be based on the upper extremity and will include various types of exercises and the primary affected November muscles in the upper extremity. It is planned that the exercises will be accompanied by a physiotherapist 2 days a week, with a total of 16 sessions for 8 weeks. It is planned that there will be a total of 8-10 exercises in 10 repetitions in the exercise program. The total length of the exercise session will be 30 minutes. It is planned that the same physiotherapist will be one-on-one with the patient from the beginning to the end of the exercises.
  Groups: non-operative conservative treatment; scapulothoracic arthrodesis
Diagnostic Test: Results of assessment — The total follow-up period of participants included in intervention programs will be 8 weeks. Evaluations will be evaluated by physiotherapist before and at the end of treatment.

SUMMARY:
Facioscapulohumeral Muscular Dystrophy (FSHD) is one of the most common forms of muscular dystrophy, characterized by pronounced skeletal weakness and with a broad spectrum of diseases. It is a hereditary disease seen in 3-5/100,000 of society, usually starting with weakness in the facial and shoulder muscles and progressing to the trunk, pelvis and leg muscles, giving symptoms in the twenties. In FSHD, which shows slow progression and can lead to loss of ambulation ability in about 20% of patients, patients may have difficulty performing activities above shoulder level with the influence of the periscapular area.

The goal of FSHD treatment is to improve muscle strength and/or function. Treatments include medical, conservative and surgical methods. The aim of surgical methods is to improve shoulder function and prevent pain caused by the movements of the scapula. The publications on physiotherapy interventions and aerobic exercise are available as conservative treatment. In patients diagnosed with FSHD, conservative treatment is frequently used to improve muscle strength, regulate function and improve the quality of life of patients.

Patients with FSHD use their affected upper extremities asymmetrically, which leads to the development of restrictive compensation mechanisms in the development of symmetrical postural control. Postural control deficits may occur due to limited use of the affected scapula in individuals with FSHD. Accordingly, in cases with FSHD, there is the use of atypical movements for balance and mobility. It is not yet known whether people with FSHD really have poorer dynamic stability during self-initiated whole-body movements such as walking, and at what stage of the disease these difficulties arise.

Accordingly, the aim of this study was to examine the effects of rehabilitation approaches applied to the upper limb on upper limb function, balance and walking in patients with FSHD.

H1: Within the group of patients with FSHD patients underwent surgery arthrodesis surgery scapulothoracic applied to pre-treatment with the parameters of the rehabilitation program for the evaluation of upper limb functionality after applying the upper extremities, postural control and gait parameters examined, there is statistical difference between the groups.

DETAILED DESCRIPTION:
Voluntary participants who have been diagnosed with FSHD and agreed to voluntary health subjects will be included in the study. Signed voluntary consent will be obtained from participants. Participants will be divided into tree groups. One group will include patients who have undergone scapulothoracic arthrodesis surgery, while the other group will include patients who have not undergone surgery and control group will include participants who have agree to participate the study. A progressive rehabilitation program for the upper extremities will be applied to patients in a group of individuals who have undergone and have not undergone surgery. Both groups will undergo some outcome measures to assess their upper extremity function, balance and walking.

ELIGIBILITY:
Inclusion Criteria:

* Individuals to be included in all groups 18-50 years
* Score between 0.5 and 3.5 according to CSS (Clinical Severity Score) of the cases to be included in the intervention groups.
* Be rated between 3-5 according to FAS (functional ambulation scale) of the cases to be included in intervention groups
* For patients who will be included in the intervention group who have undergone surgery, bilateral scapulothoracic arthrodesis surgery within 3 months at the earliest
* Individuals who will be included in the control group consisting of healthy individuals have not undergone any orthopedic surgery

Exclusion Criteria:

* Having received regular physiotherapy for 1 month, at least 2 days a week in the last 6 months
* Presence of additional neurological problem/problems
* Presence of any other upper limb problem/problems and surgery
* Presence of lower limb problems/problems that can cause balance and walking problems
* Having undergone Spinal fusion surgery
* Having lower back pain described 6 and above according to VAS (Visual Analog Scale) in intervention and control groups
* Having a level of visual and auditory problems that will prevent communication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who have been diagnosed with FSHD, patients who have undergone scapulothoracic arthrodesis, healthy people for control group
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-04-23 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
change from baseline 10 Meter Walk Test value at 8 weeks | baseline and every four weeks up to eight week
  during the test, the patient is asked to walk at a normal walking speed at a distance of 10 meters determined before the test. The time it has traveled the specified distance is recorded. It is a long-term performance test used for dynamic balance assessment.
change from baseline Gait Analyzer for walking speed at 8 weeks (m/sec) | baseline and every four weeks up to eight week
  It is a smartphone-based application for analyzing walking parameters in real time. It can measure walking speed, step time, step length, cadence and symmetry.
change from baseline Gait Analyzer for step time at 8 weeks (sec) | baseline and every four weeks up to eight week
  It is a smartphone-based application for analyzing walking parameters in real time. It can measure walking speed, step time, step length, cadence and symmetry.
change from baseline Gait Analyzer for step lenght at 8 weeks (m) | baseline and every four weeks up to eight week
  It is a smartphone-based application for analyzing walking parameters in real time. It can measure walking speed, step time, step length, cadence and symmetry.
change from baseline Gait Analyzer for cadance at 8 weeks (step/min) | baseline and every four weeks up to eight week
  It is a smartphone-based application for analyzing walking parameters in real time. It can measure walking speed, step time, step length, cadence and symmetry.
change from baseline Gait Analyzer for symmetry at 8 weeks (%) | baseline and every four weeks up to eight week
  It is a smartphone-based application for analyzing walking parameters in real time. It can measure walking speed, step time, step length, cadence and symmetry.

SECONDARY OUTCOMES:
change from baseline Timed up and Go Test at 8 weeks | baseline and every four weeks up to eight week
  The test is a measure of dynamic equilibrium. It requires individuals to get up from a chair, walk 3 feet, turn and sit. The time from the moment the individual lifts the pelvis from the chair until he or she returns with the pelvis in the chair is recorded in seconds.
change from baseline Single Leg Stance Test at 8 weeks | baseline and every four weeks up to eight week
  It is used to evaluate static posture and balance control. The patient must stand unaided on one leg from the moment the other foot leaves the ground until the foot touches the ground again or the arms are separated from the hips.
change from baseline 30 Seconds Sit Up Test at 8 weeks | baseline and every four weeks up to eight week
  It is a test that evaluates the patient's sit-up activity, lower limb strength and dynamic balance. A 30-second period is initiated when the patient cuts the contact of his pelvis from the chair in which he is sitting. He is constantly asked to sit on the chair and get up from there within 30 seconds. It is scored by counting how many repetitions the patient applies this command within 30 seconds
change from baseline Hand-Held Dynamometer values at 8 weeks | baseline and every four weeks up to eight week
  It is an efficient, objective, precise and affordable alternative to muscle strength measurement. A small portable device is held by the examiner and placed towards the patient's limb during maximum isometric contraction.
change from baseline Pedometer values at 8 weeks | baseline and every four weeks up to eight week
  It is a proven, inexpensive system that helps to measure the steps of individuals with the help of sensors attached to the ankle.
change from baseline Patient Satisfaction Questionnare at 8 weeks | every four weeks up to eight week
  It is a scale in which the fifth likert scale is used and patients report their satisfaction with the results of the treatments they receive. The points given are between -2 and +2.The higher scores indicate a better result.
Disabilities of Arm, Shoulder and Hand | baseline and every four weeks up to eight week
  It is a questionnaire that examines the patient's ability to perform certain upper extremity activities. This questionnaire is a self-report questionnaire in which patients evaluate their difficulties and situations in daily life
Berg Balance Scale | baseline and every four weeks up to eight week
  This scale evaluates the static and dynamic balance by observing the patient's performance for each instruction and giving a score between 0-4. Better scores indicate better balance.

CONTACTS AND LOCATIONS:
Overall Officials: Ipek Yeldan Karagoz, PhD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Fecek C, Emmady PD. Facioscapulohumeral Muscular Dystrophy. 2023 Jun 26. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK559028/ PMID 32644454
- [Background] Rijken NH, van Engelen BG, Weerdesteyn V, Geurts AC. Clinical Functional Capacity Testing in Patients With Facioscapulohumeral Muscular Dystrophy: Construct Validity and Interrater Reliability of Antigravity Tests. Arch Phys Med Rehabil. 2015 Dec;96(12):2201-6. doi: 10.1016/j.apmr.2015.08.429. Epub 2015 Sep 9. PMID 26363336
- [Background] Tawil R, Van Der Maarel SM. Facioscapulohumeral muscular dystrophy. Muscle Nerve. 2006 Jul;34(1):1-15. doi: 10.1002/mus.20522. PMID 16508966
- [Background] Kang PB, Morrison L, Iannaccone ST, Graham RJ, Bonnemann CG, Rutkowski A, Hornyak J, Wang CH, North K, Oskoui M, Getchius TS, Cox JA, Hagen EE, Gronseth G, Griggs RC; Guideline Development Subcommittee of the American Academy of Neurology and the Practice Issues Review Panel of the American Association of Neuromuscular & Electrodiagnostic Medicine. Evidence-based guideline summary: evaluation, diagnosis, and management of congenital muscular dystrophy: Report of the Guideline Development Subcommittee of the American Academy of Neurology and the Practice Issues Review Panel of the American Association of Neuromuscular & Electrodiagnostic Medicine. Neurology. 2015 Mar 31;84(13):1369-78. doi: 10.1212/WNL.0000000000001416. PMID 25825463
- [Background] Tawil R, Kissel JT, Heatwole C, Pandya S, Gronseth G, Benatar M; Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology; Practice Issues Review Panel of the American Association of Neuromuscular & Electrodiagnostic Medicine. Evidence-based guideline summary: Evaluation, diagnosis, and management of facioscapulohumeral muscular dystrophy: Report of the Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology and the Practice Issues Review Panel of the American Association of Neuromuscular & Electrodiagnostic Medicine. Neurology. 2015 Jul 28;85(4):357-64. doi: 10.1212/WNL.0000000000001783. PMID 26215877
- [Background] Kord D, Liu E, Horner NS, Athwal GS, Khan M, Alolabi B. Outcomes of scapulothoracic fusion in facioscapulohumeral muscular dystrophy: A systematic review. Shoulder Elbow. 2020 Apr;12(2):75-90. doi: 10.1177/1758573219866195. Epub 2019 Aug 14. PMID 32313557
- [Background] Iosa M, Mazza C, Pecoraro F, Aprile I, Ricci E, Cappozzo A. Control of the upper body movements during level walking in patients with facioscapulohumeral dystrophy. Gait Posture. 2010 Jan;31(1):68-72. doi: 10.1016/j.gaitpost.2009.08.247. Epub 2009 Sep 25. PMID 19782569
- [Background] Rijken NH, van Engelen BG, de Rooy JW, Weerdesteyn V, Geurts AC. Gait propulsion in patients with facioscapulohumeral muscular dystrophy and ankle plantarflexor weakness. Gait Posture. 2015 Feb;41(2):476-81. doi: 10.1016/j.gaitpost.2014.11.013. Epub 2014 Dec 2. PMID 25687333
- [Background] Eagle M. Report on the muscular dystrophy campaign workshop: exercise in neuromuscular diseases Newcastle, January 2002. Neuromuscul Disord. 2002 Dec;12(10):975-83. doi: 10.1016/s0960-8966(02)00136-0. No abstract available. PMID 12467755
- [Background] Statland JM, Tawil R. Risk of functional impairment in Facioscapulohumeral muscular dystrophy. Muscle Nerve. 2014 Apr;49(4):520-7. doi: 10.1002/mus.23949. Epub 2014 Feb 10. PMID 23873337